CLINICAL TRIAL: NCT04629014
Title: Prospective Multisite Study of Quality of Life in Pediatric Intestinal Failure
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Seattle Children's Hospital (Other); University of Alabama at Birmingham (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Washington University School of Medicine (Other); University of Michigan (Other); Duke Health (Other); University of Texas Southwestern Medical Center (Other); Alberta Children's Hospital (Other); British Columbia Children's Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Biren Modi, Surgical Director, Center for Advanced Intestinal Rehabilitation, Boston Children's Hospital
Other Study IDs: P00032389
Record Dates: First submitted 2020-10-29; First posted 2020-11-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Intestinal Failure
Keywords: intestinal failure; short bowel syndrome; short gut syndrome; parenteral nutrition; specialized nutrition
MeSH Terms: conditions — Intestinal Failure; Short Bowel Syndrome; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study proposes to quantify and describe the quality of life of children with intestinal failure, and to identify the medical and socio-economic factors that impact this quality of life, using data from multiple multidisciplinary intestinal failure centers across the United States and Canada specializing in the care of these participants.

DETAILED DESCRIPTION:
Health related quality of life is becoming an increasingly important topic as medical advancements continue to increase life expectancies in various illnesses. Quality of life (QoL) encompasses the physical, psychological, and social well-being of a person. Studies focusing on health related QoL show that providers have a limited understanding of the QoL of their patients, demonstrating a need for further research. Mortality rates in pediatric intestinal failure (PIF) have significantly dropped over the past 3-4 decades and long-term morbidity rather than survival has come into focus as the outcome of interest. However, there remains a significant knowledge gap regarding the specific factors that contribute to QoL among PIF patients and their families. Insight into the challenges these patients face can promote enhanced support services and psycho-education for caregivers of these children as well as help to tailor medical and surgical treatment with a focus on improved QoL. Due to the rare nature of PIF, and despite a recent bloom in multidisciplinary PIF centers, experience is limited in individual centers and a multi-site study with a robust and diverse patient population is optimal to study QoL in pediatric intestinal failure.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be followed in a participating institution's intestinal rehabilitation program
* Participants will have a diagnosis of intestinal failure due to functional or structural intestinal dysfunction with current or prior history of specialized nutritional support (parenteral nutrition requirement for 60 out of 74 consecutive days)
* Participants will be age 6 months to 25 years old.
* Parents/caregivers must be able to complete questionnaire without assistance.
* English or Spanish speaking

Exclusion Criteria:

* Participants aged less than 6 months or greater than 25 years will not be included in this study
* Participants will not be enrolled less than 3 months from index admission or initial outpatient evaluation
* Participants will not be enrolled less than 1 month from inpatient admission (any admission greater than 24 hours in duration)
* Participants will not be enrolled less than 1 month from any operative intervention requiring general anesthesia.
* Primary language other than English or Spanish.
* Participants who have a currently functional small bowel, liver/small bowel or multivisceral transplant
* While other major co-morbidities may be excluded at a later time during data analysis, or may be analyzed as a specific sub-group, they will not be excluded outright. For example, participants with global developmental delay may have parent surveys only, and therefore would need to be excluded from paired analysis of proxy vs. participant perception of HRQOL

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be children with a specific diagnosis of intestinal failure as determined by parenteral nutrition dependence at any point in their history for more than 60 out of 74 consecutive days who are managed at one of the intestinal rehabilitation programs located at the study participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (hrQOL) | Baseline
  hrQOL as determined by PedsQL Generic Core at time of enrollment and corrected for time from onset of disease
Health-related quality of life (hrQOL) Change over time | Trend over 5 years
  hrQOL as determined by PedsQL Generic Core, assessed annually, looking at trend in change over 5 years of assessment and corrected for time from onset of disease
Disease-specific Health-related quality of life (hrQOL) | Baseline
  Disease-specific hrQOL as determined by PedsQL GI Symptoms Scale at time of enrollment and corrected for time from onset of disease
Disease-specific Health-related quality of life (hrQOL) | Trend over 5 years
  Disease-specific hrQOL as determined by PedsQL GI Symptoms Scale, assessed annually, looking at trend in change over 5 years of assessment and corrected for time from onset of disease

SECONDARY OUTCOMES:
Family Impact | Baseline
  Family impact as determined by the PedsQL Family Impact Module
Family Impact | Trend over 5 years
  Family impact as assessed by the PedsQL Family Impact Module, assessed annually, looking at trend in change over 5 years of assessment and corrected for time from onset of disease

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Javid, MD, Principal Investigator — Seattle Children's Hospital; Biren P Modi, MD MPH, Principal Investigator — Boston Children's Hospital
Locations (11):
- United States (8):
  - Children's of Alabama, Birmingham, Alabama
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Duke Children's Hospital, Durham, North Carolina
  - Dallas Children's Hospital, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diamond IR, de Silva N, Pencharz PB, Kim JH, Wales PW; Group for the Improvement of Intestinal Function and Treatment. Neonatal short bowel syndrome outcomes after the establishment of the first Canadian multidisciplinary intestinal rehabilitation program: preliminary experience. J Pediatr Surg. 2007 May;42(5):806-11. doi: 10.1016/j.jpedsurg.2006.12.033. PMID 17502188
- [Background] Javid PJ, Malone FR, Reyes J, Healey PJ, Horslen SP. The experience of a regional pediatric intestinal failure program: Successful outcomes from intestinal rehabilitation. Am J Surg. 2010 May;199(5):676-9. doi: 10.1016/j.amjsurg.2010.01.013. PMID 20466115
- [Background] Modi BP, Langer M, Ching YA, Valim C, Waterford SD, Iglesias J, Duro D, Lo C, Jaksic T, Duggan C. Improved survival in a multidisciplinary short bowel syndrome program. J Pediatr Surg. 2008 Jan;43(1):20-4. doi: 10.1016/j.jpedsurg.2007.09.014. PMID 18206449
- [Background] Mutanen A, Kosola S, Merras-Salmio L, Kolho KL, Pakarinen MP. Long-term health-related quality of life of patients with pediatric onset intestinal failure. J Pediatr Surg. 2015 Nov;50(11):1854-8. doi: 10.1016/j.jpedsurg.2015.05.012. Epub 2015 Jun 3. PMID 26078213
- [Background] Norsa L, Artru S, Lambe C, Talbotec C, Pigneur B, Ruemmele F, Colomb V, Capito C, Chardot C, Lacaille F, Goulet O. Long term outcomes of intestinal rehabilitation in children with neonatal very short bowel syndrome: Parenteral nutrition or intestinal transplantation. Clin Nutr. 2019 Apr;38(2):926-933. doi: 10.1016/j.clnu.2018.02.004. Epub 2018 Feb 15. PMID 29478887
- [Background] Sanchez SE, McAteer JP, Goldin AB, Horslen S, Huebner CE, Javid PJ. Health-related quality of life in children with intestinal failure. J Pediatr Gastroenterol Nutr. 2013 Sep;57(3):330-4. doi: 10.1097/MPG.0b013e3182999961. PMID 23648789
- [Background] Varni JW, Limbers CA, Burwinkle TM. Impaired health-related quality of life in children and adolescents with chronic conditions: a comparative analysis of 10 disease clusters and 33 disease categories/severities utilizing the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jul 16;5:43. doi: 10.1186/1477-7525-5-43. PMID 17634123
- [Derived] Modi BP, Piper HG, Belza C, Staffa S, Arnold MA, Boctor DL, Channabasappa N, Cohran VC, Galloway DP, Sudan D, Wales PW, Warner BW, Murtadi G, Javid PJ. Health-Related Quality of Life in Pediatric Intestinal Failure from Infancy to Adolescence: An International, Multi-Center Evaluation. J Pediatr. 2025 Jul;282:114566. doi: 10.1016/j.jpeds.2025.114566. Epub 2025 Mar 28. PMID 40158842